CLINICAL TRIAL: NCT01309386
Title: A Randomized, Open-Label, Parallel-Arm, Optimal Dose-Titration, Multicenter Study to Evaluate the Safety and Efficacy of Oral JNS024 Extended-Release (ER) in Japanese Subjects Treated With Around-the-Clock Opioid Analgesics for Their Moderate to Severe Chronic Malignant Tumor- Related Cancer Pain
Brief Title: A Safety and Efficacy Study of Oral Tapentadol Extended-Release in Japanese Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017326; JNS024ER-JPN-C03
Record Dates: First submitted 2011-02-17; First posted 2011-03-07 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-02

CONDITIONS: Neoplasms
Keywords: Tapentadol; Tumor related pain; Opioid; Cancer related pain; Morphine
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol ER (Experimental): Tapentadol extended-release (ER) (JNS024ER) oral tablets 100 to 400 milligram (mg) daily for 8 weeks (maximum dose could be up to 500 mg daily), as per Investigator's discretion.
  Interventions: Drug: Tapentadol ER
- Morphine SR (Active Comparator): Morphine sustained-release (SR) oral tablets 30 to 120 mg daily for 8 weeks (maximum dose could be up to 140 mg daily), as per Investigator's discretion.
  Interventions: Drug: Morphine SR

INTERVENTIONS:
Drug: Tapentadol ER — Tapentadol ER 100 to 400 milligram (mg) orally daily for 8 weeks (maximum up to 500 mg daily), as per Investigator's discretion.
  Arms: Tapentadol ER
Drug: Morphine SR — Morphine SR 30 to 120 mg orally daily for 8 weeks (maximum up to 140 mg daily), as per Investigator's discretion.
  Arms: Morphine SR

SUMMARY:
The purpose of this study is to evaluate the conversion rate based on the number of participants achieving pain control and safety within 1 week after switching the opioid (morphine-like medications) analgesics (drug used to control pain), when tapentadol extended-release (ER) (JNS024ER) is orally administered to participants treated with around-the-clock opioid analgesics, for their moderate to severe (very serious, life threatening) chronic (lasting a long time) malignant (cancerous) tumor-related (a mass in a specific area) cancer (abnormal tissue that grows and spreads in the body) pain.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), parallel-arm (participants receive 1 of 2 possible interventions during the same time frame throughout the study), optimal dose-titration, multicenter (when more than one hospital or medical school team work on a medical research study) study evaluating the conversion rate based on the number of participants achieving pain control and safety within 1 week after switching from an ongoing around-the-clock opioid analgesic (morphine sustained-release [SR], oxycodone controlled-release, or fentanyl transdermal) to tapentadol ER or morphine SR, for their moderate to severe chronic, malignant tumor-related cancer pain. The study consists of 2 periods: 1 to 2 week screening period, followed by 8-week open-label treatment period. During the study period, participants will be hospitalized or outpatient. However, it is preferable to be hospitalized 1 week before and 1 week after to evaluate efficacy before and after switching opioids for securing participants' safety. At Day 1, participants will receive either tapentadol ER or morphine SR twice daily. During the treatment period, the dose of the study drug will be titrated to the participant's optimal dose. The participants will receive either tapentadol ER or morphine SR twice daily for 8 weeks. The maximum dose allowed for tapentadol ER will be 500 milligram (mg) daily or morphine SR 140 mg daily throughout the study. Efficacy is primarily evaluated using pain intensity score on an 11 point Numerical Rating Scale (an 11-point NRS is used to measure the pain level where 0=no pain to 10=pain as bad as you can imagine). Participants' safety will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented clinical diagnosis (determination of the cause of a medical problem) of any type of cancer (abnormal tissue that grows and spreads in the body)
* Participants with mean 24-hour Numerical Rating Scale (NRS) score (11-point NRS used to measure the pain level for the past 24-hours where 0=no pain to 10=pain as bad as you can imagine) during 3 days (Day -4 to Day -2) before randomization (study drug assigned by chance) less than 4.0
* Women must be post-menopausal, surgically sterile, or before entry and throughout the study practicing an effective method of birth control
* Participants using immediate-release (IR) morphine hydrochloride (HCl) or oxycodone HCl hydrate as rescue medication (rescue medications are medicines that may be administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation) for breakthrough pain
* Participants treated with around-the-clock opioid (morphine-like medications) therapy for moderate to severe (very serious, life threatening) chronic (lasting a long time), malignant (cancerous) tumor-related (a mass in a specific area) cancer (abnormal tissue that grows and spreads in the body) pain using one of the following opioid analgesics (drug used to control pain) before randomization: morphine SR tablet less than or equal to 120 milligram (mg) per day, oxycodone hydrochloride controlled release (CR) tablet: 15 mg to 80 mg per day, durotep MT (fentanyl transdermal [through the skin] matrix) patch less than or equal to 8.4 mg per patch, fentos tape less than or equal to 4 mg per tape, or oneduro patch less than or equal to 3.4 mg per patch

Exclusion Criteria:

* Participants with complicated uncontrolled/clinically significant arrhythmia (uneven heart beat)
* Participants who had received rescue doses 3 times or more daily within 3 days (Day -4 to Day -2) before the randomization
* History of surgery intended for the cure of the primary disease or for the treatment of cancer pain within 28 days before screening
* Participants who had application of radiotherapy (treatment of cancer using x-rays), nerve block, or stimulation analgesia within 7 days before screening
* Participants with known allergies (over sensitivity to a substance), hypersensitivity, or intolerance to opioid analgesics or its excipients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (22):
- Japan (22):
  - Chiba
  - Hamamatsu
  - Ibaraki
  - Kanagawa
  - Katsushika-ku
  - Kobe
  - Kumamoto
  - Matsumoto
  - Matsuyama
  - Nagasaki
  - Nagoya
  - Nishinomiya
  - Ohmura
  - Ohta
  - Osaka
  - Saga
  - Sapporo
  - Tokyo
  - Toyama
  - Toyohashi
  - Utsunomiya
  - Yokohama

REFERENCES:
- [Derived] Imanaka K, Tominaga Y, Etropolski M, Ohashi H, Hirose K, Matsumura T. Ready conversion of patients with well-controlled, moderate to severe, chronic malignant tumor-related pain on other opioids to tapentadol extended release. Clin Drug Investig. 2014 Jul;34(7):501-11. doi: 10.1007/s40261-014-0204-3. PMID 24906437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tapentadol ER | Morphine SR
Started | 50 | 50
Completed | 28 | 29
Not Completed | 22 | 21
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Progressive disease | 9 | 11
Not completed — Physician Decision | 1 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Adverse Event | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol ER | Morphine SR | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Number; unit: Participants]
  Less than 65 years | 23 (8.5) | 25 (9.97) | 48
  More than or equal to 65 years | 27 | 25 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Pain Control
Description: Pain control was considered to be achieved for participants who met both of the following criteria for any consecutive 3 days during the first week of treatment period: a) Change from baseline of mean 24 hour numerical rating scale (NRS) (an 11-point NRS is used to measure the pain level where 0=no pain to 10=pain as bad as you can imagine) score less than +1.5, and b) when the frequency of rescue medication was twice or less per day.
Time Frame: Week 1
Population: Full analysis set (FAS) population included all participants who were randomly assigned, received at least 1 dose of study drug and had post-baseline efficacy data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Percentage of Participants | 84.0 [70.89 to 92.83] | 98.0 [89.35 to 99.95]

2. Secondary Outcome: Change From Baseline in Numerical Rating Scale (NRS) at Week 1, 2, 3, 4, 5, 6, 7 and 8
Description: Average pain intensity was assessed using an 11-point NRS to measure the pain level for the past 24-hours where 0=no pain to 10=pain as bad as you can imagine.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
Population: Full analysis set (FAS) population included all participants who were randomly assigned, received at least 1 dose of study drug and had post-baseline efficacy data. Here 'n' signifies those participants evaluable for this measure at the specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Unit on scale
  Change at Week 1 (n = 50, 50) | 0.4 (0.92) | -0.2 (0.84)
  Change at Week 2 (n = 45, 44) | 0.3 (1.11) | -0.3 (0.75)
  Change at Week 3 (n= 41, 41) | 0.1 (0.90) | -0.1 (1.03)
  Change at Week 4 (n = 38, 37) | 0.1 (0.90) | -0.3 (0.95)
  Change at Week 5 (n = 36, 34) | 0.1 (0.92) | -0.1 (1.22)
  Change at Week 6 (n = 36, 32) | 0.2 (0.97) | 0.1 (1.43)
  Change at Week 7 (n = 34, 29) | 0.1 (1.00) | 0.1 (1.05)
  Change at Week 8 (n = 29, 29) | 0.0 (0.92) | 0.0 (1.21)

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to Lack of Efficacy
Description: Number of participants who discontinued the treatment due to lack of efficacy were assessed throughout the study.
Time Frame: Baseline up to Week 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Participants | 3 | 1

4. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGIC)
Description: The PGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the participant's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved".
Time Frame: Week 1, 4 and 8
Population: Full analysis set (FAS) population; here 'N' signifies those participants evaluable for this outcome measure and 'n' signifies those participants evaluable for this measure at the specified time point for each arm group, respectively.
Measure: Number; unit: Participants
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 48 | 48
Participants
  Week 1 (very much improved) (n=48,48) | 1 | 2
  Week 1 (much improved) (n=48,48) | 1 | 4
  Week 1 (minimally improved) (n=48,48) | 11 | 7
  Week 1 (not changed) (n=48,48) | 24 | 29
  Week 1 (minimally worse) (n=48,48) | 9 | 6
  Week 1 (much worse) (n=48,48) | 2 | 0
  Week 1 (very much worse) (n=48,48) | 0 | 0
  Week 4 (very much improved) (n=37,37) | 1 | 3
  Week 4 (much improved) (n=37,37) | 2 | 5
  Week 4 (minimally improved) (n=37,37) | 9 | 7
  Week 4 (not changed) (n=37,37) | 22 | 19
  Week 4 (minimally worse) (n=37,37) | 3 | 3
  Week 4 (much worse) (n=37,37) | 0 | 0
  Week 4 (very much worse) (n=37,37) | 0 | 0
  Week 8 (very much improved) (n=28,28) | 0 | 3
  Week 8 (much improved) (n=28,28) | 3 | 2
  Week 8 (minimally improved) (n=28,28) | 8 | 4
  Week 8 (not changed) (n=28,28) | 15 | 13
  Week 8 (minimally worse) (n=28,28) | 2 | 4
  Week 8 (much worse) (n=28,28) | 0 | 2
  Week 8 (very much worse) (n=28,28) | 0 | 0

5. Secondary Outcome: Total Number of Days of Rescue Medication Over Time
Description: Total number of days of rescue medication over time were assessed. Rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Supplemental analgesics (drug used to control pain) were used as rescue medication.
Time Frame: Baseline up to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Days | 15.9 (19.58) | 9.2 (12.76)

6. Secondary Outcome: Number of Doses of Rescue Medication Over Time
Description: Number of doses of rescue medication over time were assessed. Rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Supplemental analgesics (drug used to control pain) were used as rescue medication.
Time Frame: Baseline up to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Morphine-equivalent doses
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Morphine-equivalent doses | 0.7 (0.89) | 0.4 (0.53)

7. Secondary Outcome: Average Change From Baseline in Amount of Rescue Medication Over Time
Description: Rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Supplemental analgesics (drug used to control pain) were used as rescue medication. Average amount was the averages of all doses recorded during the baseline period or during each week (Week 1, 2, 3, 4, 5, 6, 7 and 8).
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram (mg)
Arm/Group | Tapentadol ER | Morphine SR
Number analyzed (Participants) | 50 | 50
Milligram (mg) | 3.02 (8.303) | -0.15 (5.038)

ADVERSE EVENTS:
Arm/Group | Tapentadol ER | Morphine SR
Serious Adverse Events (participants affected / at risk) | 16/50 | 16/50
Other Adverse Events (participants affected / at risk) | 43/50 | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=50) | Morphine SR (N=50)
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Disease progression (General disorders) | 10 | 10
Condition aggravated (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=50) | Morphine SR (N=50)
Nasopharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Delirium (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1
Senile psychosis (Psychiatric disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Somnolence (Nervous system disorders) | 8 | 10
Headache (Nervous system disorders) | 1 | 4
Dizziness (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Slow response to stimuli (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 7 | 7
Vomiting (Gastrointestinal disorders) | 2 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urobilinuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 4
Disease progression (General disorders) | 9 | 8
Chest pain (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Catheter site swelling (General disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 1
Glucose urine present (Investigations) | 0 | 2
Neutrophil count increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 1
Protein urine present (Investigations) | 0 | 2
Blood urea increased (Investigations) | 0 | 1
Differential white blood cell count abnormal (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Malaise (General disorders) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.